CLINICAL TRIAL: NCT04975568
Title: Effectiveness of Therapeutic Exercise Controlled Through App Adding Face-to-face Supervision Executed by Physical Therapist in the Subacute and Chronic Low Back Pain
Brief Title: Effectiveness of Therapeutic Exercise App Adding a Face-to-face Physical Therapist in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI 19/514-E
Record Dates: First submitted 2021-06-10; First posted 2021-07-23 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain
Keywords: Physiotherapy; Mobile Applications; Therapeutic Exercise
MeSH Terms: conditions — Low Back Pain | interventions — Amyloid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercise Controlled Through App With face-to-face (Experimental): 3 months treatment using app for HTEP and 6 people therapeutic exercise group every 15 days
  Interventions: Other: App and face-to-face physical therapy; Other: App physical therapy
- Therapeutic Exercise Controlled Through App (Active Comparator): 3 months treatment using app for HTEP
  Interventions: Other: App physical therapy

INTERVENTIONS:
Other: App and face-to-face physical therapy — Patients will use an app with health tests, general information about the study, personalized HTEP based in McGill's Program after their evaluations, and several online materials related with healthcare and healthy habits linked to social media sites. During the app used they will have 6 face-to-face sessions in 6 people groups with a physical Therapist in a 3 months period
  Arms: Therapeutic Exercise Controlled Through App With face-to-face
Other: App physical therapy — Patients will use an app with health tests, general information about the study, personalized HTEP based in McGill's Program after their evaluations, and several online materials related with healthcare and healthy habits linked to social media sites.

SUMMARY:
Low Back Pain (LBP) is one of the most usual illness in our society. Therapeutic Exercise (TE) has been shown the most effective and cheaper treatment in patients suffering LBP, but the lack of engagement to the therapeutic exercise programs is related with later acute LBP and chronic situations, despite symptoms slightly improve.

The value of personalized therapeutic exercised programs in patients suffering LBP has been shown nowadays, improving symptomatology and quality of life.

New technologies help patients to engage more in treatment, while time that health education make people "active patients".

The aim of the study is to evaluate the effectiveness of a Home Therapeutic Exercise Program (HTEP) based in an app with McGill's exercised adding 6 face-to-face sessions every 15 days with a physical therapist .

DETAILED DESCRIPTION:
INTRODUCTION

Low back pain is defined as pain and discomfort, localized below the costal margin and above the inferior gluteal folds, with or without leg pain . Sub-acute low back pain as low back pain persisting between 6 and 12 weeks; chronic low back pain as low back pain persisting for 12 weeks or more. It is not usual define specific causes of LBP, no more than 15 % patients have a define cause. Non-specific low back pain is defined as low back pain not attributed to recognizable, known specific pathology (e.g. infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome or cauda equina syndrome).

LBP is one of main world health problems, 23.9 % world citizens suffer LBP over a month in their life. World aging foresee this percentage will increase more in women from 40 to 80 years old. In 2017 LBP was an important men and women chronic health problem in Spain, the second cause more important in women with 23.5 % Spanish women suffering it and the third one in men with 15.8 % Spanish men suffering it. LBP is also the most important cause of work absenteeism with general back pain and migraine.

LBP is related with sedentary lifestyle. Recurrent low back pain is usual. There are several studies searching LBP's risks and LBP's risks factors but they did not show a clear reason.

Studies about app beef up treatment engagement and treatment effectiveness. Last studies about engagement and health improvement using app had shown positive results in diabetes patients, hypertension patients, heart pathology or daily pain management without help (for example Keele Pain Recorder app).

There is a wide and proven evidence of the improvement in symptomatology using app to prescribe exercise in patients suffering LBP according to Sunil et al papers (aerobic daily programs plus 7 specific exercise towards LBP treatment), proposing health mobile apps as an important tool to chronic pathologies.

But in front of the positive situation of a better engagement, app use has a couple of limitations as the reinforcement that a face-to-face control provides ant the information that a specialist health professional can add to the app mobile development to improve the final results.

JUSTIFICATION

LBP is one of the most important health problems of our society. The present study postulates the possible link between technology and real treatment, proposing a HTEP created to non-specific LBP with an app, using McGill's Big Three exercise as the base of the program.

McGill's Big Three Exercise are 3 basic and low complexity exercises to treat any patient who is suffering non-specific low back pain, that had shown a real effectiveness in order to reduce pain intensity and to get better functionality. McGill proposed 3-exercise warm up before the Big Three "Curl up", "Side Bridge" and "Bird Dog" that had to be executed in an isometric contraction. Maximal muscular contraction had to be under 8 seconds, because longer contraction would reduce effectiveness as McGill showed in one of his studies.

The study will propose an individualized McGill Program using an app as support to the two arms of the study, and the main difference will be that experimental group will have a face-to-face control every 15 days and the control group will work only with the app.

App development has the supervision or three specialized physical therapists in LBP.

HYPOTHESIS

The addition of 6 face-to-face sessions executed by physical therapist to the personalized HTEP provided by the app is more effective at improving pain intensity, functionality, quality of life and treatment engagement in patients suffering non-specific LBP.

OBJECTIVES

General:

Evaluate the effectiveness of adding face-to-face supervision sessions executed by Physical Therapist to a HTEP with an app in people suffering non-specific LBP.

Specifics

1. Evaluate the effectiveness of adding face-to-face supervision sessions executed by Physical Therapist to a HTEP with an app in people suffering non-specific LBP reducing pain intensity measured by PI-NRS.
2. Evaluate the effectiveness of adding face-to-face supervision sessions executed by Physical Therapist to a HTEP with an app in people suffering non-specific LBP improving functionality measured by Oswestry scale.
3. Evaluate the effectiveness of adding face-to-face supervision sessions executed by Physical Therapist to a HTEP with an app in people suffering non-specific LBP improving life quality of life measured by SF-12 scale.
4. Evaluate patient satisfaction degree of a semi presential treatment measured by PSQ.
5. Evaluate the effectiveness of adding face-to-face supervision sessions executed by Physical Therapist to a HTEP with an app in people suffering non-specific LBP improving engagement treatment analyzing app database.

METHODOLOGY

Type of study: randomized and controlled pilot study, in a two arms study with parallel interventions the experimental one and the control one. The study will blind randomization, patient assessment and data analysis. Patient randomization will take place at "Universidad Complutense de Madrid" using random permutations model of Moses and Oakford. Study characteristics itself prevent their blinded application cause:

* Evaluators (baseline, intervention, and post-intervention) will be different professionals that physical therapist will provide face-to-face sessions, and they will ignore in which group patients are in.
* Physical therapist that provide face-to-face sessions will not have any evaluation data.

This study will assure blinded randomization assessment, recruiters and evaluators of assessment group of each patient.

Location: Universidad Complutense de Madrid. Study Subjects: 90 patients suffering non-specific LBP

Sample size: This study has a paper published in 2018 as reference and the standard deviation was 2 in pain measure variable.

Accepting an alpha risk of 0.5 and a beta risk of 0.2 in a two-sided test, 90 subjects (45 in the control group and 45 in the experimental group) are necessary to recognize as statistically significant a difference greater than or equal to 1.5 units. The standard deviation is assumed to be 2, and it has been anticipated a drop-out rate of 10 %.

Data collection and analysis. Before starting the study, all patients will be asked to sign an informed consent in the first session where it will take place the initial assessment including the collection of patient data records and the booklet of questionnaires and clinical measurements using the app.

The patient will receive weekly 3 sessions of his personalized HTEP and experimental group will receive also 6 group session every 15 days t controlled by a physical therapist.

1. At first session, before treatment, variables PI-NRS, SF-12 and Oswestry variables will be measured.
2. 2 weeks after baseline, before treatment, PI-NRS variable will be measured.
3. 4 weeks after baseline, before treatment, SF-12 and Oswestry variables will be measured.
4. 6 weeks after baseline, before treatment, PI-NRS variable will be measured.
5. 8 weeks after baseline, before treatment, SF-12 and Oswestry variables will be measured.
6. 10 weeks after baseline, before treatment, PI-NRS variable will be measured.
7. 12 weeks after baseline the patient will be re-evaluated. PI-NRS, Oswestry, SF-12, PSQ and engagement variables will be measure The following week to the end of treatment, the patient will be re-evaluated.

The statistical analysis will be performed using SPSS 22.0 program (IBM statistical software).

The average and the standard deviation of quantitative variables will be calculated for the descriptive analysis of the sample. In non-normal distributions the nonparametric sum of the ranges of Wilcoxon and Chi Square test will be performed, as well as the homogeneity in baseline will be displayed by overlapping confidence intervals.

For the comparative analysis, developed according to the intention to treat:

1. A MANOVA (ANOVA for repeated measures) test should be carry out to evaluate the interaction between levels of inter - subject factor (treatment) and the intra- subject (main variables response in time) to be interpreted in case it is significant.
2. To confirm whether this interaction effect is significant, pairwise comparisons will be made of the inter-subjects factor levels (treatment) for each level of main response variables over time using the Bonferroni method.

Limitations of the study and measures taken to reduce them.

Masking: The nature of the applied treatments prevents masking therapists and patients. This limitation is inherent to the type of treatment evaluated and common with other forms of treatment with similar characteristics, in which therapist should inevitably know the type of treatment that is applied.

However, this limitation does not prevent the controlled clinical trials carried out on these technologies from being of higher methodological quality. Thus, in this study, randomization of patients will be blind, allocation of the random sequence, the assessment of patient evolution and analysis of results.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 65 years old.
* Suffering low back pain.
* In a subacute and chronic phase

Exclusion Criteria:

* Non signature of the informed consent
* Red Flags are risk factors detected in low back pain patients' past medical history and symptomatology and are associated with a higher risk of serious disorders causing low back pain compared to patients without these characteristics.
* Yellow Flags are psychosocial factors that increase the risk of developing, or perpetuating chronic pain and long-term disability (including) work-loss associated with low back pain.
* Pregnancy and lactation
* Serious trauma or back surgery before the study
* Illness or dysfunction of balance
* Visual dysfunction.
* Neurological illness, dysfunction or pain.
* Inability to stand up and sit without help
* Inability to read, understand and complete questionnaires, read and understand a brochure, or understand and follow verbal instructions (e.g. Illiteracy, dementia or blindness) or read, understand and use an app

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with improve intensity of Low Back pain based in Pain Intensity- Numerical Rating Scale | 12 weeks treatment
  Intensity of low back pain (measured by Pain Intensity- Numerical Rating Scale ( PI-NRS)) at rest. It will be valued three times with 1 min between the three valuations. 1 item, minimum value 0 and maximum value 10, and 10 is the worse value and the average will be recorded.

SECONDARY OUTCOMES:
Number of participants with improve degree of Low Back pain disability based in Oswestry test | At baseline, 4 weeks treatment, 8 weeks treatmentment,12 weeks treatment and 2 months post-treatment
  Low Back pain disability (measured by Oswestry test). 10 items and 10 points each item, the minimun value is 0 the maximum is 100, and 100 is the worse outcome
Number of participants with improve degree of quality of life based in Spanish version of the Short Form Health Survey | At baseline, 4 weeks treatment, 8 weeks treatmentment,12 weeks treatment and 2 months post-treatment
  Quality of life (measured by a previously validated Spanish version of the Short Form Health Survey (SF-12)) 12 items, the minimun value is 12 the maximum is 55, and 55 is the worse outcome
Level of physical therapy intervention satisfaction based in Spanish version of the Patient Satisfaction Questionnaire | 12 weeks treatment
  Satisfaction (measured by a previously validated Spanish version of the Patient Satisfaction Questionnaire (PSQ)) 13 items, the minimun value is 13 the maximum is 78, and 78 is the worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jose Javier Lopez Marcos, Master, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Jose Javier López Marcos, Madrid, Spain

REFERENCES:
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Background] Mesas AE, Gonzalez AD, Mesas CE, de Andrade SM, Magro IS, del Llano J. The association of chronic neck pain, low back pain, and migraine with absenteeism due to health problems in Spanish workers. Spine (Phila Pa 1976). 2014 Jul 1;39(15):1243-53. doi: 10.1097/BRS.0000000000000387. PMID 24825151
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Lotzke H, Jakobsson M, Gutke A, Hagstromer M, Brisby H, Hagg O, Smeets R, Lundberg M. Patients with severe low back pain exhibit a low level of physical activity before lumbar fusion surgery: a cross-sectional study. BMC Musculoskelet Disord. 2018 Oct 11;19(1):365. doi: 10.1186/s12891-018-2274-5. PMID 30305065
- [Background] da Silva T, Mills K, Brown BT, Herbert RD, Maher CG, Hancock MJ. Risk of Recurrence of Low Back Pain: A Systematic Review. J Orthop Sports Phys Ther. 2017 May;47(5):305-313. doi: 10.2519/jospt.2017.7415. Epub 2017 Mar 29. PMID 28355981
- [Background] Hanney WJ, Masaracchio M, Liu X, Kolber MJ. The Influence of Physical Therapy Guideline Adherence on Healthcare Utilization and Costs among Patients with Low Back Pain: A Systematic Review of the Literature. PLoS One. 2016 Jun 10;11(6):e0156799. doi: 10.1371/journal.pone.0156799. eCollection 2016. PMID 27285608
- [Background] Kleinman NJ, Shah A, Shah S, Phatak S, Viswanathan V. Improved Medication Adherence and Frequency of Blood Glucose Self-Testing Using an m-Health Platform Versus Usual Care in a Multisite Randomized Clinical Trial Among People with Type 2 Diabetes in India. Telemed J E Health. 2017 Sep;23(9):733-740. doi: 10.1089/tmj.2016.0265. Epub 2017 Mar 6. PMID 28328396
- [Background] Chao DY, Lin TM, Ma WY. Enhanced Self-Efficacy and Behavioral Changes Among Patients With Diabetes: Cloud-Based Mobile Health Platform and Mobile App Service. JMIR Diabetes. 2019 May 10;4(2):e11017. doi: 10.2196/11017. PMID 31094324
- [Background] Marquez Contreras E, Marquez Rivero S, Rodriguez Garcia E, Lopez-Garcia-Ramos L, Carlos Pastoriza Vilas J, Baldonedo Suarez A, Gracia Diez C, Gil Guillen V, Martell Claros N; Compliance Group of Spanish Society of Hypertension (SEH-LELHA). Specific hypertension smartphone application to improve medication adherence in hypertension: a cluster-randomized trial. Curr Med Res Opin. 2019 Jan;35(1):167-173. doi: 10.1080/03007995.2018.1549026. Epub 2018 Dec 5. PMID 30431384
- [Background] Santo K, Singleton A, Chow CK, Redfern J. Evaluating Reach, Acceptability, Utility, and Engagement with An App-Based Intervention to Improve Medication Adherence in Patients with Coronary Heart Disease in the MedApp-CHD Study: A Mixed-Methods Evaluation. Med Sci (Basel). 2019 Jun 4;7(6):68. doi: 10.3390/medsci7060068. PMID 31167489
- [Background] Bedson J, Hill J, White D, Chen Y, Wathall S, Dent S, Cooke K, van der Windt D. Development and validation of a pain monitoring app for patients with musculoskeletal conditions (The Keele pain recorder feasibility study). BMC Med Inform Decis Mak. 2019 Jan 25;19(1):24. doi: 10.1186/s12911-019-0741-z. PMID 30683106
- [Background] Chhabra HS, Sharma S, Verma S. Smartphone app in self-management of chronic low back pain: a randomized controlled trial. Eur Spine J. 2018 Nov;27(11):2862-2874. doi: 10.1007/s00586-018-5788-5. Epub 2018 Oct 15. PMID 30324496
- [Background] Machado GC, Pinheiro MB, Lee H, Ahmed OH, Hendrick P, Williams C, Kamper SJ. Smartphone apps for the self-management of low back pain: A systematic review. Best Pract Res Clin Rheumatol. 2016 Dec;30(6):1098-1109. doi: 10.1016/j.berh.2017.04.002. Epub 2017 May 25. PMID 29103552
- [Background] Durall CJ, Udermann BE, Johansen DR, Gibson B, Reineke DM, Reuteman P. The effects of preseason trunk muscle training on low-back pain occurrence in women collegiate gymnasts. J Strength Cond Res. 2009 Jan;23(1):86-92. doi: 10.1519/JSC.0b013e31818b93ac. PMID 19057402
- [Background] Hewett TE, Myer GD, Ford KR. Reducing knee and anterior cruciate ligament injuries among female athletes: a systematic review of neuromuscular training interventions. J Knee Surg. 2005 Jan;18(1):82-8. doi: 10.1055/s-0030-1248163. PMID 15742602
- [Background] McGill SM, Hughson RL, Parks K. Lumbar erector spinae oxygenation during prolonged contractions: implications for prolonged work. Ergonomics. 2000 Apr;43(4):486-93. doi: 10.1080/001401300184369. PMID 10801082
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- See also: Chapter 4. European guidelines for the management of chronic nonspecific low back pain. European Spine Journal : Official Publication of the European Spine Society — https://doi.org/10.1007/s00586-006-1072-1
- See also: Instituto nacional de estadística. Mujeres y Hombres en España. — https://www.ine.es/ss/Satellite?L=es_ES&c=INESeccion_C&cid=1259926692949&p=1254735110672&pagename=ProductosYServicios%2FPYSLayout&param1=PYSDetalle&param3=1259924822888
- See also: Instituto nacional de estadística — https://www.ine.es/jaxi/Datos.htm?path=/t00/ICV/dim3/l0/&file=33302.px
- See also: Adaptación y validación de un cuestionario para medir la satisfacción del tratamiento de fisioterapia en atención primaria — https://dialnet.unirioja.es/servlet/tesis?codigo=156680